CLINICAL TRIAL: NCT00764218
Title: Cardiovascular Phenotype Study in Patients With Obstructive Sleep Apnea Syndrome : Role of Hypertension
Brief Title: Cardiovascular Phenotype Study in Patients With Obstructive Sleep Apnea Syndrome
Acronym: SAS-HTA
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: BAGUET Jean-Philippe, PhD, University Hospital Grenoble
Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DGS2001/0398
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2008-10-01 (Estimated); Status verified 2001-01

CONDITIONS: Obstructive Sleep Apnea Syndrome; Hypertension
Keywords: Obstructive sleep apnea syndrome; Hypertension; Cardiovascular phenotype
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- SAS+HTA+ (Experimental): Obstructive sleep apnea syndrome and hypertension
  Interventions: Device: Positive airway pressure treatment
- SAS+HTA- (Experimental): non hypertensive patients with obstructive sleep apnea syndrome
  Interventions: Device: Positive airway pressure treatment
- SAS-HTA+ (Experimental): hypertensive patients without obstructive sleep apnea syndrome
  Interventions: Other: No positive airway pressure treatment
- SAS-HTA- (Experimental): non hypertensive patients without obstructive sleep apnea syndrome
  Interventions: Other: No positive airway pressure treatment

INTERVENTIONS:
Device: Positive airway pressure treatment — Positive airway pressure treatment as long as necessary
  Other Names: CPAP treatment
  Arms: SAS+HTA+; SAS+HTA-
Other: No positive airway pressure treatment — No treatment
  Other Names: No CPAP treatment
  Arms: SAS-HTA+; SAS-HTA-

SUMMARY:
Patients with obstructive sleep apnea syndrome have permanent variations of their hemodynamic parameters during the night : heart rate, arterial blood pressure, cardiac output. This is due to the repetition of respiratory events (obstructive apnea and hypopnea) leading to frequent micro-arousals. These disorders have several consequences : hypertension, NO-dependent vasodilatation impairment, baroreceptor reflex impairment, insulin resistance and other cardiovascular impairments.

DETAILED DESCRIPTION:
Objective of the study is to characterize the cardiovascular phenotype of patients with obstructive sleep apnea syndrome, relative to the presence of hypertension or not. Hypertension should not have been previously treated. 2 groups of apneic patients (SAS+HTA+ and SAS+HTA-) will be compared together, referred to group of non apneic but hypertensive patients (SAS-HTA+) and non apneic / non hypertensive patients (SAS-HTA-).

Apneic and hypertensive patients may have a sympathetic nervous system activation and a much more important vascular and baroreceptor reflex impairment, than non apneic but hypertensive patients.

During the study, a second visit as control will be done for apneic patients only, 3 to 6 months after SAS treatment setting.

ELIGIBILITY:
Inclusion Criteria:

* patients with or without obstructive sleep apnea syndrome (AHI > 15)
* patients with or without hypertension

Exclusion Criteria:

* known or expected secondary hypertension
* pathologies with consequences on arterial blood pressure regulation: Parkinson's disease, patients with renal or cardiac graft, severe heart failure
* drugs with consequences on arterial blood pressure regulation : vasoconstrictors, vasodilatators, béta-agonists, antagonists, nitrites, theophylline, dipyridamol, sildenafil, immunosuppressors, IMAO, neuroleptics, tricyclic antidepressants, corticoids or long-term oral (>10 days) non steroidal anti-inflammatory drugs, oestroprogestative treatments
* atrial fibrillation, frequent extrasystoles (> or = to 10/minute)
* bedridden patients
* night shift workers
* surgical or carotid stenting history
* subjects unwilling or unable to provide written, signed and dated informed consent
* patient previously treated for obstructive sleep apnea syndrome (positive airway pressure, forward mandible prosthesis, maxillofacial surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-03; Primary Completion 2003-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
cardiovascular phenotype study in patients with non treated obstructive sleep apnea syndrome | 6 years

SECONDARY OUTCOMES:
characterization of arterial blood pressure, sympathetic activity, functional and morphological cardiovascular modifications. Effect of a treatment of obstructive sleep apnea syndrome on those different parameters. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe JB BAGUET, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Cardiology and hypertension service, Grenoble, Isère, France

REFERENCES:
- [Background] Pankow W, Nabe B, Lies A, Becker H, Kohler U, Kohl FV, Lohmann FW. Influence of sleep apnea on 24-hour blood pressure. Chest. 1997 Nov 5;112(5):1253-8. doi: 10.1378/chest.112.5.1253. PMID 9367465
- [Background] Portaluppi F, Provini F, Cortelli P, Plazzi G, Bertozzi N, Manfredini R, Fersini C, Lugaresi E. Undiagnosed sleep-disordered breathing among male nondippers with essential hypertension. J Hypertens. 1997 Nov;15(11):1227-33. doi: 10.1097/00004872-199715110-00006. PMID 9383171
- [Background] Calver A, Collier J, Moncada S, Vallance P. Effect of local intra-arterial NG-monomethyl-L-arginine in patients with hypertension: the nitric oxide dilator mechanism appears abnormal. J Hypertens. 1992 Sep;10(9):1025-31. PMID 1328361
- [Background] Strohl KP, Novak RD, Singer W, Cahan C, Boehm KD, Denko CW, Hoffstem VS. Insulin levels, blood pressure and sleep apnea. Sleep. 1994 Oct;17(7):614-8. doi: 10.1093/sleep/17.7.614. PMID 7846459
- [Background] Landsberg L. Hyperinsulinemia: possible role in obesity-induced hypertension. Hypertension. 1992 Jan;19(1 Suppl):I61-6. doi: 10.1161/01.hyp.19.1_suppl.i61. PMID 1730456
- [Background] Carlson JT, Hedner JA, Sellgren J, Elam M, Wallin BG. Depressed baroreflex sensitivity in patients with obstructive sleep apnea. Am J Respir Crit Care Med. 1996 Nov;154(5):1490-6. doi: 10.1164/ajrccm.154.5.8912770.
- [Background] Peppard PE, Young T, Palta M, Skatrud J. Prospective study of the association between sleep-disordered breathing and hypertension. N Engl J Med. 2000 May 11;342(19):1378-84. doi: 10.1056/NEJM200005113421901. PMID 10805822
- [Background] Nieto FJ, Young TB, Lind BK, Shahar E, Samet JM, Redline S, D'Agostino RB, Newman AB, Lebowitz MD, Pickering TG. Association of sleep-disordered breathing, sleep apnea, and hypertension in a large community-based study. Sleep Heart Health Study. JAMA. 2000 Apr 12;283(14):1829-36. doi: 10.1001/jama.283.14.1829. PMID 10770144
- [Background] Baguet JP, Mallion JM, Moreau-Gaudry A, Noirclerc M, Peoc'h M, Siche JP. Relationships between cardiovascular remodelling and the pulse pressure in never treated hypertension. J Hum Hypertens. 2000 Jan;14(1):23-30. doi: 10.1038/sj.jhh.1000933. PMID 10673727
- [Derived] Baguet JP, Barone-Rochette G, Levy P, Vautrin E, Pierre H, Ormezzano O, Pepin JL. Left ventricular diastolic dysfunction is linked to severity of obstructive sleep apnoea. Eur Respir J. 2010 Dec;36(6):1323-9. doi: 10.1183/09031936.00165709. Epub 2010 Jun 18. PMID 20562120
- [Derived] Baguet JP, Nadra M, Barone-Rochette G, Ormezzano O, Pierre H, Pepin JL. Early cardiovascular abnormalities in newly diagnosed obstructive sleep apnea. Vasc Health Risk Manag. 2009;5:1063-73. doi: 10.2147/vhrm.s8300. Epub 2009 Dec 29. PMID 20057899